CLINICAL TRIAL: NCT04369573
Title: Early Intra-aortic Balloon Pump Placement in Acute Decompensated Heart Failure Complicated by Cardiogenic Shock: a Randomized Clinical Trial
Brief Title: Study on Early Intra-aortic Balloon Pump Placement in Acute Decompensated Heart Failure Complicated by Cardiogenic Shock
Acronym: Altshock-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because the Data Safety Monitoring Board after the interim analisys concluded that the experimental treatment is not proviiding any minimal full benefit compared to the contrtol. They then reccomended to stop the trial due to futility
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S_21_08_19_3263
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cardiogenic Shock
Keywords: Acute decompensated heart failure; cardiogenic shock; intra-aortic balloon pump
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Drug Implants; Standard of Care

STUDY DESIGN:
Intervention Model Description: Multicentre Prospective Controlled Randomized Trial in patients with ADHF complicated by CS. Patients will be randomized 1:1 to early IABP versus standard of care. Early IABP will be defined as IABP implantation for CS patients within 6 hours since CS symptoms onset.
Masking Description: Open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intra-aortic balloon pump (IABP) implantation (Active Comparator): IABP implantation within 6 hours since cardiogenic shock symptoms onset
  Interventions: Combination Product: Early intra-aortic balloon pump (IABP) implantation
- Standard of care as vasoactive agent (Other): Any agent (inotropes and vasopressors) will be allowed. However, the following guide is provided to increase uniformity: 1) vasopressors allowed will be either epinephrine or norepinephrine; 2) as inotropic agent milrinone or dobutamine or levosimendan could be used; 3) dopamine will be allowed in association with milrinone or dobutamine or levosimendan; 4) the maximum inotropic score allowed will be 20
  Interventions: Other: Standard of care as vasoactive agent

INTERVENTIONS:
Combination Product: Early intra-aortic balloon pump (IABP) implantation — IABP implantation within 6 hours since cardiogenic shock symptoms onset
  Arms: Early intra-aortic balloon pump (IABP) implantation
Other: Standard of care as vasoactive agent — Any agent (inotropes and vasopressors) will be allowed. However, the following guide is provided to increase uniformity: 1) vasopressors allowed will be either epinephrine or norepinephrine; 2) as inotropic agent milrinone or dobutamine or levosimendan could be used; 3) dopamine will be allowed in association with milrinone or dobutamine or levosimendan; 4) the maximum inotropic score allowed will be 20.
  Arms: Standard of care as vasoactive agent

SUMMARY:
The aim of the study is to demonstrate the superiority of early intra-aortic balloon pump implantation at admission over local clinical practice (pharmacological only) in acute decompensated heart failure patients with cardiogenic shock, with respect to 60-day survival or successful bridge to heart replacement therapies (heart transplant or Left Ventricular Assist Device implantation).

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is the most severe form of acute heart failure, with in-hospital mortality up to 50%. Failure to improve mortality has been reported, despite observed improvements in hemodynamics. Previous studies on CS have almost exclusively been focused on CS following an acute coronary syndrome (ACS). Chronic heart failure patients with acute decompensation (ADHF) and CS represent a unique physiologic phenotype compared with ACS patients, which may lead to a differential response to device therapy. Recent evidences emphasize that intra-aortic balloon pump (IABP) is not recommended for patients with ACS-related CS, but it is associated with a high likelihood of bridge to durable Left Ventricular Assist Device or heart transplant without the need for escalation to more potent temporary mechanical circulatory support devices, when implanted in ADHF patients. Data retrieved from the available literature in the setting of patients with CS not related to ACS are poor even in large, well-reported registries.

Accordingly, Altshock-2 trial has been designed to test the superiority of early IABP implantation at admission over local clinical practice (pharmacological only) in ADHF patients with CS, with respect to 60-day survival or successful bridge to heart replacement therapies

ELIGIBILITY:
INCLUSION CRITERIA

* Age ≥ 18 and < 75, men and women;
* need of vasoactive agents to maintain SBP > 90 mmHg or MAP > 60 mmHg.
* Left ventricle systolic function ≤35%
* SCAI B-D according to CSWG definition (JACC 2022)

EXCLUSION CRITERIA

* septic shock with evident septic focus;
* severe peripheral vascular disease
* CS secondary to cardiac and non-cardiac surgery;
* Acute myocardial infarction within 1 month;
* Suspected or documented myocarditis
* Pulmonary embolism
* Chronic end-stage organ dysfunction that would preclude heart transplant/durable VAD
* ominous prognosis (life expectancy < 1 year);
* any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
* pregnant, lactating or women planning pregnancy during the course of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Successful bridge to heart replacement therapies, namely heart transplantation or left ventricular assist device implantation | 60 days
  Number of participants to heart transplant or Left Ventricular Assist Device implantation
Survival | 60 days
  Rate

SECONDARY OUTCOMES:
Renal replacement therapy, namely any need of replacement of kidney function due to renal failure by means of the following techniques: continuous hemofiltration and hemodialysis, intermittent hemodialysis, and peritoneal dialysis | 60 days
  Number of participants who need a renal replacement therapy among the two groups (early IABP vs standard)
Maximum inotropic score among the two groups | Through study completion, an avererage of 30 days
  To compare maximum inotropic score among the two groups (early IABP vs standard).
  IS (mcg/kg/min) = [dopamine, dobutamine + 100 x (norepinephrine+epinephrine) +15 x IPDE-3 +10for levosimendan] (Reference: Int J Artif Organs. 2016 Feb;39(2):94-7)
Maximum duration of inotropic/vasopressor therapy among the two groups | Through study completion, an avererage of 30 days
  To compare maximum duration of inotropic/vasopressor therapy among the two groups (early IABP vs standard)
Maximum sequential organ failure assessment (SOFA) | Through study completion, an avererage of 30 days
  To compare maximum sequential organ failure assessment (SOFA)
early IABP vs standard | 60 days
  To compare 60-day overall survival among the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morici N, Sacco A, Frea S, Rota M, Villanova L, Gravinese C, Dini CS, D'Ettore N, Maj G, De Lio G, Potena L, Valente S, Sabatino M, Viola G, Garatti L, Tavecchia GA, Bertoldi L, Oliva F, Kapur NK, Tavazzi G, De Ferrari GM, Pappalardo F; Altshock-2 Investigators. Early Intra-Aortic Balloon Support for Heart Failure-Related Cardiogenic Shock: A Randomized Clinical Trial. J Am Coll Cardiol. 2025 Apr 29;85(16):1587-1597. doi: 10.1016/j.jacc.2025.03.003. Epub 2025 Mar 30. PMID 40162941